CLINICAL TRIAL: NCT01174693
Title: Comparison of Triflusal and Clopidogrel Effect in Secondary Prevention of Stroke Based on the Cytochrome P450 2C19 Genotyping
Brief Title: Comparison of Triflusal and Clopidogrel in Secondary Prevention of Stroke Based on the Genotyping
Acronym: MAESTRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Collaborators: Myung In Pharmaceutical Company (Unknown); Yonsei University (Other)
Responsible Party: Principal Investigator, KyungYul Lee, MD, PhD, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAESTRO-001
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Cerebral Infarction
Keywords: prospective; randomized; open label; multi-center; double-blind for CYP2C19 genotypes
MeSH Terms: conditions — Cerebral Infarction | interventions — triflusal; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel (Active Comparator): Plavix® 75mg tablet, 75mg once daily, Mode of administration: oral, Duration: from randomization to 31 December 2014
  Interventions: Drug: Clopidogrel
- Triflusal (Experimental): Disgre® 150mg or 300mg capsule, 300mg bid, Mode of administration: oral, Duration: from randomization to 31 December 2014
  Interventions: Drug: Triflusal

INTERVENTIONS:
Drug: Triflusal — Dose: 150mg or 300mg capsule, 300mg bid, Mode of administration: oral, Duration: from randomization to 31 December 2014
  Other Names: Disgren®
  Arms: Triflusal
Drug: Clopidogrel — Dose: 75mg tablet, 75mg once daily, Mode of administration: oral, Duration: from randomization to 31 December 2014
  Other Names: Plavix®
  Arms: Clopidogrel

SUMMARY:
The purpose of this study is to compare the preventive effect of stroke between triflusal and clopidogrel in ischemic stroke patient based on the cytochrome P450 2C19 (CYP2C19) polymorphism.

DETAILED DESCRIPTION:
Clopidogrel has anti-platelet activity by irreversible inhibition of the P2Y12 platelet receptor. Clopidogrel must be converted into an active metabolite in order to show anti-platelet activity. Hepatic CYP2C19 enzyme is one of the key hepatic enzymes which convert clopidogrel into active metabolite and its genetic polymorphism is related to clopidogrel resistance. CYP2C19 poor or intermediate metabolizer groups show reduced anti-platelet activity of clopidogrel compared to extensive metabolizer group.

This study is designed to prove the superiority of the triflusal in preventing recurrent stroke over the clopidogrel in ischemic stroke patient with poor or intermediate metabolizer of CYP2C19 polymorphism. Also we plan to prove that clopidogrel resistance is related to CYP2C19 polymorphism by comparing the ischemic preventive effect of clopidogrel between groups of different CYP2C19 polymorphism.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have non-cardiogenic ischemic stroke of TOAST classification within 30 days prior to screening
2. ≥ 20 years of age; adult, at the date of signing the informed consent
3. Written informed consent

Exclusion Criteria:

1. History for bleeding tendency or recent major bleeding within 2 weeks
2. Chronic liver disease (ALT > 100 IU/L or AST > 100 IU/L) or renal dysfunction (creatinine > 4.0 mg/dl)
3. Thrombocytopenia (platelet < 100,000mm3)
4. Any contraindication of antiplatelet agent
5. Severe congestive heart failure
6. Patients who need to take anticoagulants or two or more antiplatelet agents
7. Severe concomitant disease with the expected survival less than 2 years
8. Pregnant or nursing
9. Any drug clinical trials within 30 days of signing the informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 795 (Actual)
Dates: Start 2010-03; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Time to first recurrent stroke | 2.8 to 4 years
  The study will finish at least 2 years after the recruit of 1080th patients. Until the finish, patients will continuously take study medications and visit every 3months at the study site.
  We will measure primary outcome during the follow-up period (minimum 2.8 years to maximum 4 years - maximum time is determined by estimated enrollment time period of 2.8 years).

SECONDARY OUTCOMES:
Time to first of composite cardiovascular events, MI or coronary artery revascularization and ischemic stroke | 2.8 to 4 years
  The study will finish at least 2 years after the recruit of 1080th patients. Until the finish, patients will continuously take study medications and visit every 3months at the study site.
  We will measure secondary outcomes during the follow-up period (minimum 2.8 years to maximum 4 years - maximum time is determined by estimated enrollment time period of 2.8 years).

CONTACTS AND LOCATIONS:
Overall Officials: KyungYul Lee, MD, PhD, Principal Investigator — Gangnam Severance Hospital
Locations (18):
- South Korea (18):
  - Department of Neurology, Wonju Christian Hospital, Yonei University Wonju College of Medicine, Wŏnju, Gangwon-do
  - Department of Neurology, National Health Insurance Corporation Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Department of Neurology, CHA Bundang Medical Center, CHA University School of Medicine, Seongnam-si, Gyeonggi-do
  - Changwon Fatima Hospital, Changwon, Gyeongsangnam-do
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Department of Neurology, Konyang University Hospital, Daejeon
  - Department of Neurology, Chosun University Hospital, Gwangju
  - Department of Neurology, National Medical Center, Seoul
  - Department of Neurology, Severance Hospital, Yonsei University College of Medicine, Seoul
  - KyungHee University Medical Center, Seoul
  - Department of Neurology, Kyung Hee University Hospital at Gangdong, Seoul
  - Department of Neurology, Gangnam Severance Hospital, Yonsei Univ. College of Medicine, Seoul
  - Korea University Anam Hospital, Seoul
  - Department of Neurology, Sanggye Paik Hospital, Inje University College of Medicine, Seoul
  - Department of Neurology, Korea University Guro Hospital, Seoul
  - Department of Neurology, Ewha Womans University Mokdong Hospital, Seoul

REFERENCES:
- [Derived] Han SW, Kim YJ, Ahn SH, Seo WK, Yu S, Oh SH, Kim YN, Lee KY; MAESTRO Study Investigators. Protocol for the comparison of triflusal and clopidogrel in secondary prevention of stroke based on cytochrome P450 2C19 genotyping (MASETRO study): A multicenter, randomized, open-label, parallel-group trial. Int J Stroke. 2016 Jun;11(4):485-91. doi: 10.1177/1747493015620804. Epub 2016 Jan 5. PMID 26763917